CLINICAL TRIAL: NCT06998251
Title: In-depth Analysis of the Immune Responses in the Upper Respiratory Tract in Older Adults Infected or Colonized With Streptococcus Pneumoniae (Spn)
Acronym: NoseSpnElderly
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Arnaud Didierlaurent, Professor, University of Geneva, Switzerland
Other Study IDs: 2024-01135
Record Dates: First submitted 2025-03-28; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Pneumococcal Infections; Respiratory Syncytial Virus (RSV) Infection; Influenza Infection
MeSH Terms: conditions — Pneumococcal Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasal cells, nasal lining fluid, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Spn patients: Patients hospitalized with community-acquired pneumonia due to a Streptococcus pneumoniae infection
- Flu/RSV patients: Patients hospitalized with flu-like symptoms and a laboratory-confirmed influenza or RSV infection
- Asymptomatic Spn carriers: Healthy people screened for asymptomatic carriage of Streptococcus pneumoniae

SUMMARY:
The NoseSpn-Elderly study aims at characterizing the immune response in the upper respiratory tract in adults aged 60 and over diagnosed with a pneumonia due to a Streptococcus pneumoniae (Spn) infection. The immune response during the acute phase of the infection and after recovery will be compared to the immune response of asymptomatic Spn carriers as well as to the immune response of patients diagnosed with a viral respiratory infection (flu or respiratory syncytial virus (RSV)).

The primary objective of this observational study is to quantify the inflammatory response in the nasal cavity and to correlate it with bacterial/viral load and with clinical parameters. The study also aims to compare the inflammatory response measured in the nose to that measured in the blood.

Participants will have two study visits including a blood draw, several nasal samplings (nasal lining fluid and nasal cells) and a saliva sampling, one within 72 hours of their hospital admission and another one month later. Nasal lining fluid and saliva will be obtained every two or three days until discharge from the hospital or resolution of symptoms. During those visits, questions regarding symptoms will be asked.

ELIGIBILITY:
Inclusion criteria:

* Aged 60-85 years
* Able to provide informed consent either independently or by a legal representative
* Group 1 (Spn pneumonia patients): clinical and/or radiological signs of pneumonia
* Group 1 (Spn pneumonia patients): positive Spn urinary antigen and/or blood culture and/or positive sputum test.
* Group 2 (viral respiratory infection patients): clinical signs of a respiratory infection
* Group 2 (viral respiratory infection patients): positive test for influenza or RSV
* Group 3 (asymptomatic Spn-carriers): healthy without clinical signs of infection and no lower respiratory symptoms within the last month.

Exclusion criteria:

* Immunosuppression,
* Use of inhalation and/or nasal steroids the last month
* Intubation or under invasive mechanical ventilation
* Long-term antibiotic treatment prior to disease onset

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 and group 2 participants will be recruited among patients hospitalized or consulting the emergencies at the Geneva University Hospitals (HUG). Group 3 participants will be recruited among participants of other HUG studies involving healthy adults as well as from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pro-inflammatory cytokine levels in nasal fluid by a multiplex assay | 1 month

SECONDARY OUTCOMES:
Phenotypes and frequencies of immune in nasal cavity and in blood cells by flow cytometry | 1 month
Antibody titers in nasal cavity and blood by antigen-specific ELISA | 1 month
Bacterial load and viral load in nasal cavity by specific qPCR assay | 1 month
Levels of serum cytokines by multiplex assay | 1 month
Clinical outcome measure 1: pneumonia diagnostic | 1 month
  Probability of diagnosis of pneumonia (on a 3-Likert scale: low, intermediate and high level of probability)
Clinical outcome measure 2: CURB65 severity score | 1 month
Clinical outcome measure 3: nature and severity of symptoms (CAP score) | 1 month
Clinical outcome measure 4: number of days with fever | 1 month
Clinical outcome measure 5: number of days with oxygen | 1 month
Clinical outcome measure 6: highest FiO2 | 1 month
Clinical outcome measure 7: cardiac complication | 1 month
Clinical outcome measure 8: secondary bacterial infection | 1 month
  Only for group 2 patients (viral infection)
Clinical outcome measure 9: transfer to ICU or IMCU | 1 month
Clinical outcome measure 10: length of stay in intensive care | 1 month
Clinical outcome measure 11: intubation or mechanical ventilation | 1 month
Clinical outcome measure 12: transfer to rehabilitation or institutionalization | 1 month
Clinical outcome measure 13: mortality | 1 month
Clinical outcome measure 14: rehospitalization | 1 month
Clinical outcome measure 15: medical consultation for a respiratory disease | 1 month
Clinical outcome measure 16: new prescription of antibiotics or corticosteroids | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Didierlaurent, PhD, Principal Investigator — University of Geneva; Virginie Prendki, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland